CLINICAL TRIAL: NCT04609059
Title: First-in-Patient Study for Sing le Dose of M201-A Hydrochloride Injection in Japanese Patients With Paroxysmal Atrial Fibrillation
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kitasato University (Other)
Collaborators: Aetas Pharma Co. Ltd. (Industry)
Responsible Party: Principal Investigator, Yuji KUMAGAI, Yuji KUMAGAI, Professor, Kitasato University, Kitasato University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M201-A-CT-002
Record Dates: First submitted 2020-09-16; First posted 2020-10-30 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- M201-A Injection (Experimental): Active Substance: M201-A Route of administration: continuous intravenous injection
  Interventions: Drug: M201-A Injection
- Placebo (Placebo Comparator): Saline Placebo for M201-A Route of administration: continuous intravenous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: M201-A Injection — Active Substance: M201-A Route of administration: continuous intravenous injection
  Step 1: Continuous Intravenous Injection administered with single dose of M201-A hydrochloride or placebo 0.4 mg/kg in 50 mL, controlled with a syringe driver at a rate of 2.5 mL/min for 20 minutes Step 2: Continuous Intravenous Injection administered with single dose of M201-A hydrochloride or placebo 0.6 mg/kg in 50 mL, controlled with a syringe driver at a rate of 2.5 mL/min for 20 minutes (Based on recommendations of an independent data monitoring committee; data and safety monitoring board, it will be decided that dosage is 0.20 mg/kg or 0.40 mg/kg. If appropriate, Step 2 will not be conducted.)
  Arms: M201-A Injection
Drug: Placebo — Saline Placebo: M201-A Placebo Route of administration: continuous intravenous injection
  Step 1: Continuous Intravenous Injection administered with single dose of M201-A hydrochloride or placebo 0.4 mg/kg in 50 mL, controlled with a syringe driver at a rate of 2.5 mL/min for 20 minutes Step 2: Continuous Intravenous Injection administered with single dose of M201-A hydrochloride or placebo 0.6 mg/kg in 50 mL, controlled with a syringe driver at a rate of 2.5 mL/min for 20 minutes (Based on recommendations of an independent data monitoring committee; data and safety monitoring board, it will be decided that dosage is 0.20 mg/kg or 0.40 mg/kg. If appropriate, Step 2 will not be conducted.)
  Arms: Placebo

SUMMARY:
First-in-Patient Study for sing le dose of M201-A hydrochloride injection in Japanese patients with paroxysmal atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* (1) Japanese (male, female) adult with symptomatic paroxysmal atrial fibrillation (AF)
* Written informed consent must be obtained on a voluntary basis before any assessment is performed.

  (2) Age: 20 to less than 85 years of age (3) Weight: 40 kilograms(kg) or more BMI: 18.5 to less than 28.0 on screening examination(screening) (4) Past AF History: Event(s) as symptomatic AF with (at least) 2 hours or more AF lasting has (have) occurred at least once or more a half year (6 months) prior to the screening.

  (5) Occurrence time of the latest AF: Record(s) of the patient portable electrocardiograph shows evidence to support that the latest AF has occurred within 3 hours to less than 3 days (72 hours) prior to an administration of the investigational product.

  (6) The AF lasting prior to the administration: 12 lead electrocardiogram just prior to the administration shows that AF has not stopped.

  (7) Excluded medication: Based on propositions of a principal investigator or a co-investigator(s), a patient can consent for discontinuation of below antiarrhythmic agents (the Vaughan-Williams classification) for at least 7 days after administration since an advanced registration. Nonetheless, if a period between the advanced registration and the administration is less than 7 days, it should be confirmed those agent has unadministered during 7 days prior to the administration.

[Vaughan-Williams classification] Antiarrhythmic drug group I Antiarrhythmic drug group III Antiarrhythmic drug group IV Bepridil (8) Excluded administration of amiodarone: It should be confirmed that amiodarone hydrochloride is not unadministered within one (1) year before the screening.

Exclusion Criteria:

* (1) Heart failure (NYHA II, III, IV). Excluding palpitations induced by atrial fibrillation (AF) (2) Any atrioventricular block of first, second or third degree at the time of sinus rhythm (3) Any risk factor leads to Torsades de Pointes (TdP)

  1. [0]: 440 ms or more in standard 12-lead electrocardiogram at the time of sinus rhythm within 3 months prior to administration
  2. Hypokalemia or suspected to be hypokalemia:

     One or more of serum potassium levels, obtained at any time during 6 months in advance of administration including pre-administration examination, has been 3.6 [1]/L or less.
  3. Hypomagnesemia or suspected be hypomagnesemia: One or more of serum magnesium levels, obtained at any time during 6 months in advance of administration including pre-administration examination, has been 1.8 mg/dL or less.
  4. T-wave abnormality of electrocardiogram at the time of sinus rhythm
  5. Past medical history as fainting; syncope with unknown etiology or complicating illness.
  6. Past own medical history or family medical history as long QT syndrome (4) Severe heart hypertrophy; Cardiomegaly: Septal Thickness of cardiac ultrasound has been exceeded over 15 mm.

     (5) Left atrial dimension (parasternal long-axis view) of cardiac ultrasound has been exceeded over 45 mm.

Ages: 20 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety Assessment | throughout the study duration(up to day7)
  Safety investigation based on combined Investigator examination, Adverse Events (particulary, incidence of abnormal laboratory tests,abnormal vital sings,abnormal 12-lead ECG, abnormal 24-hour Holter ECG)
Arrest of atrial fibrillation (AF) | throughout the study duration(Within 2 hours)
  Ratio of arrested AF* in administered subjects within 2 hours after administration (*Restoration of sinus rhythm should be kept at least one(1) minute or more.)

CONTACTS AND LOCATIONS:
Locations (5):
- Japan (5):
  - Koga general Hospital, Koga, Ibaraki
  - Kitasato University Hospital, Sagamihara, Kanagawa
  - Sendai Cardiovascular Center, Sendai, Miyagi
  - Dokkyo Medical University Saitama Medical Center, Koshigaya, Saitama
  - Yamanashi Prefectural Central Hospital, Kofu, Yamanashi